CLINICAL TRIAL: NCT01886352
Title: Intraperitoneal Atomization of Levobupivacaine During Gynaecological Laparoscopic Procedures ; Impact on Pain, Opioid Use and Length of Recovery Room Stay (IPLA).
Acronym: IPLA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/089
Record Dates: First submitted 2013-06-07; First posted 2013-06-25 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Pain, Postoperative
Keywords: laparoscopic; pain
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Infiltration of portal sites with 0,5% levobupivacaine. (Active Comparator): The first group of patients will receive the standard treatment (paracetamol, diclofenac and an opioid if necessary) with infiltration of the portal sites with the local anesthetic ( 0.5% levobupivacaine).
  Interventions: Drug: Standard Injection of Levobupivacaine in portal sites.
- Additional injection of 0.5% levobupivacaine via a trocar (Experimental): The second group of patients will receive the standard of care, with infiltration of the portal sites with the local anesthetic ( 0.5% levobupivacaine) and additional injection of the local anesthetic ( 0.5% levobupivacaine, non -diluted) in the peritoneal cavity via a trocar both at the beginning and the end of the surgery.
  Interventions: Drug: Standard Injection of Levobupivacaine in portal sites.; Drug: Additional injection of 0,5% levobupivacaine.
- Additional intraperitoneal atomization of levobupivacaine. (Experimental): The third group of patients will receive the standard of care, with infiltration of the portal sites with the local anesthetic ( 0.5% levobupivacaine) and additional intraperitoneal atomization of the local anesthetic.
  Interventions: Drug: Standard Injection of Levobupivacaine in portal sites.; Drug: Intraperitoneal atomization of levobupivacaine.

INTERVENTIONS:
Drug: Standard Injection of Levobupivacaine in portal sites. — All port sites will be injected with 0.1ml/kg levobupivacaine at the end of surgery, after trocar removal.
Drug: Additional injection of 0,5% levobupivacaine. — Immediately following insufflation 0.15ml/kg levobupivacaine will be injected in the peritoneal cavity via a trocar. At the end of the surgery, this process will be repeated with the same dose at 0.15ml/kg.
  Arms: Additional injection of 0.5% levobupivacaine via a trocar
Drug: Intraperitoneal atomization of levobupivacaine. — Immediately following insufflation the Optispray® surgical spray device will be inserted into the abdomen and directed towards the diaphragms, dome of inflated abdomen, bowel peritoneum and surgical dissection site and the study drug will be delivered as an atomized spray in the following volumes:
  1. Each subdiaphragmatic area 0.05 ml/kg
  2. Dome of abdomen then settling onto bowel 0.05 ml/kg
  3. Surgical dissection site 0.05 ml/kg
  4. At the end of the surgery - this process will be repeated with the same doses at 0.15 ml/kg.
  Arms: Additional intraperitoneal atomization of levobupivacaine.

SUMMARY:
In this study, we will compare 3 treatments. The first group of patients will receive the standard treatment (paracetamol, diclofenac and an opioid if necessary) with infiltration of the portal sites with the local anesthetic ( 0.5% levobupivacaine) . The second group of patients will receive the standard of care, with infiltration of the portal sites with the local anesthetic ( 0.5% levobupivacaine) and additional injection of the local anesthetic ( 0.5% levobupivacaine, non -diluted) in the peritoneal cavity via a trocar both at the beginning and the end of the surgery . The third group of patients will receive the standard of care, with infiltration of the portal sites with the local anesthetic ( 0.5% levobupivacaine) and additional intraperitoneal atomization of the local anesthetic. We will use non-diluted 0.5% levobupivacaine delivered directly onto the target sites both at the beginning and the end of surgery. The drug will be delivered using OptiSpray® surgical spray device, an inexpensive delivery system that will direct a fine mist of drug directly to the areas of the peritoneal cavity that are theoretically the cause of post-op pain (diaphragms, peritoneal abdominal surface, surgical dissection site).

Our primary goal is to assess the efficacy of intraperitoneal atomization of levobupivacaine in reducing postoperative pain and of opioid requirements in patients undergoing gynecological laparoscopic procedures in one-day surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are planned for gynaecological laparoscopic interventions on an ambulatory basis.

Exclusion Criteria:

* Less than 18 year old.
* Weight less than 50 kg and more than 80 kg.
* Pregnant.
* Prisoners;
* Allergic to topical anesthetics (Amides specifically).
* Allergic to Opioids as a class.
* Currently or within the last 30 days been prescribed an opiate medication.
* Chronic pain syndrome.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-06-26 (Actual); Primary Completion 2014-06-13 (Actual); Study Completion 2018-12-03 (Actual)

PRIMARY OUTCOMES:
Post-operative pain intensity after laparoscopic gynaecological surgery in 1-day hospital setting. | Participants will be followed for the duration of hospital stay, an expected average of 1 day.
  Pain evaluation will be done using an 11-point numeric rating scale (0 = no pain, 10 = worst pain possible).
Post-operative shoulder pain after laparoscopic gynecological procedure in 1-day hospital setting. | Participants will be followed for the duration of hospital stay, an expected average of 1 day.
  Pain evaluation will be done using an 11-point numeric rating scale (0 = no pain, 10 = worst pain possible).

SECONDARY OUTCOMES:
Post-operative opioid analgesic requirements after laparoscopic gynaecological surgery. | Participants will be followed for the duration of hospital stay, an expected average of 1 day.
  Piritramide 0,05 mg/kg
Post-operative pain intensity after laparoscopic gynaecological surgery from hospital discharge until 24 hrs post-operatively. | Patients will be followed until 24 hours post-operatively.
  Patients will be asked to evaluate their pain at 6 hrs, 12 hrs, 18 hrs and 24 hrs post-operatively using an 11-point numeric rating scale (0=no pain and 10= worse pain possible) and report it by telephone.
Post-operative shoulder pain after laparoscopic gynecological surgery from hospital discharge until 24 hrs post-operatively. | Patients will be followed until 24 hours post-operatively.
  Patients will be asked to evaluate their pain at 6 hrs, 12 hrs, 18 hrs and 24 hrs post-operatively using an 11-point numeric rating scale (0=no pain and 10= worse pain possible) and report it by telephone.
Post-operative nausea and vomiting (PONV) in the first 24 hrs post-operatively, after laparoscopic gynecological surgery. | Patients will be followed until 24 hours post-operatively.
  Nausea and vomiting will be evaluated every 15' during the first 2 hrs, every 30' until hospital discharge, using a PONV verbal descriptor scale 0 to 2 points : 0=no nausea, 1=any nausea, 2 =vomiting. After discharge, patients wil be asked to evaluate PONV at 6 hrs, 12 hrs, 18 hrs and 24 hrs post-operatively and report it by telephone.
Post-operative sedation until hospital discharge, after laparoscopic gynecological surgery. | Patients will be followed up to 6 hrs post-operatively.
  Sedation will be evaluated at 0, 1, 2, 4, 6 hrs post-operatively, using the Ramsay sedation score (1= anxious and agitated, 2= cooperative, tranquil, oriented, 3=responds only to verbal commands, 4= asleep with brisk response to light stimulation, 5=asleep without response to light stimulation, 6=non-responsive).
Time until discharge from recovery room. | Up until discharge from recovery room post-operatively, probably a few hours.
  Discharge criterion: aldrete ≥ 9/10.
Time until discharge from hospital. | Patients will be followed until an estimated 24 hours post-operatively.
  Discharge criterion : modified aldrete ≥ 12/14.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Coppens, mD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

REFERENCES:
- See also: Related Info — http://www.uzgent.be